CLINICAL TRIAL: NCT07089290
Title: Effectiveness of Nurse-Led Telehealth Intervention for Hypertension Control in Nepal
Brief Title: A Study Protocol to Assess the Effectiveness of Nurse-Led Telehealth Intervention for Hypertension Control in Nepal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kathmandu University School of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bhawana Regmi, Principal Investigator, Kathmandu University School of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 369/2025
Record Dates: First submitted 2025-07-14; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Hypertension Combined Diastolic and Systolic
MeSH Terms: conditions — Systolic Murmurs

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (Active Comparator)
  Interventions: Behavioral: Nurse-led Telehealth Intervention
- Nurse-led Telehalth Intervention (Experimental)
  Interventions: Behavioral: Nurse-led Telehealth Intervention

INTERVENTIONS:
Behavioral: Nurse-led Telehealth Intervention — Control group: Patients will receive standard care as per Nepal government guidelines. This includes lifestyle counseling (salt reduction, physical activity, avoiding tobacco/alcohol), antihypertensive medications based on BP and risk profile, and follow-up every 1-3 months. BP will be recorded at 3 and 6 months by research nurses.
  Intervention group: Nurse-led telehealth care will be delivered over six months using the Intervention Mapping approach. Participants will receive initial orientation, a BP diary, and instructions to check BP at least twice weekly at nearby centers. Nurses will train local staff, and conduct teleconsultations via Viber/WhatsApp every 15 days (months 1-2) and monthly (months 3-6) covering BP review, adherence, and lifestyle advice. If <75% of BP readings meet target, nurses will consult physicians for medication adjustments. Emergency protocols will be in place. Data will be collected at baseline, 3, and 6 months.

SUMMARY:
Despite being the leading cause of cardiovascular diseases and premature death worldwide, hypertension control remains a largely unmet challenge for public health systems even in developed countries. Hypertension control in Nepal is challenging due to decreased awareness, limited access to the health facilities caused by geographical constraints and health care personnel shortage. Telehealth can help address these gaps and nurse-led telehealth can be a better option as nurses can provide timely follow up, track patients' progress and offer guidance on medication adherence and lifestyle changes which are crucial for hypertension control.

This study aims to evaluate the effectiveness of nurse-led telehealth for hypertension control among hypertensive adults in Nepal. We will use the Intervention Mapping (IM) approach to develop a theory-based and evidenced nurse-led telehealth intervention for hypertension control. Following IM, a parallel-group 1:1 randomized control trial 353 participants in each group will be used to evaluate the effectiveness of intervention. The intervention consists of regular BP monitoring, video conferencing and virtual drug adjustment. The follow up will be done in 3 and 6 months. Explanatory Sequential mixed Method will be used to assess the acceptability, appropriateness, and feasibility of adapting nurse-led telehealth for hypertension control.

Data collection will utilize a self-constructed semi-structured questionnaire, along with validated questionnaires. The collected data will be analyzed using STATA 14, contributing valuable insights into the potential impact of nurse-led telehealth interventions on increasing hypertension control.

DETAILED DESCRIPTION:
Background Hypertension (HTN) is a leading cause of cardiovascular disease and premature death worldwide. About 1.28 billion adults aged 30-79 years are estimated to have HTN; two-thirds of them are living in low and middle-income countries. Globally, 46% of adults with hypertension are estimated to be unaware that they have the condition, only 42% are diagnosed and treated, whereas only 21% have it under control. Hypertension is considered as a silent killer because most people with hypertension are not aware of the condition as it may not present warning signs and symptoms. In 2019, high systolic blood pressure was the top cause of disease burden worldwide, measured by DALYs (Disability-Adjusted Life Years). Despite the enormous burden, hypertension control remains a largely unmet challenge for public health systems, even in developed countries.

The overall prevalence of hypertension in the Asia-Pacific region ranged between 10.6% and 48.3%.6 According to a step survey 2019 in Nepal, 24.5% of adults were hypertensive, with 47.3% unaware of their condition, 29.6% of those with hypertension were receiving treatment, and among those receiving treatment, only 14.8% had their blood pressure under control. Hypertension control in Nepal faces significant challenges due to limited access to health facilities, particularly in rural areas, caused by geographical constraints and healthcare personnel shortages. Low public awareness and inadequate follow-up care further complicate the issue. Additionally, there is limited understanding of the importance of medication adherence and lifestyle modifications, hindering effective hypertension management.

Telemonitoring can help address these gaps by allowing remote monitoring of patients, enabling timely follow-up, and promoting better self-care and treatment adherence, all without the need for frequent visits to health centers. Studies in high-income countries have demonstrated that the telemonitoring of blood pressure effectively improves medication adherence and lifestyle modifications, leading to a reduction in systolic blood pressure (SBP) ranging from 5 mmHg to 32 mmHg. A study in Nepal assessed the effectiveness of mobile phone text messaging intervention where SBP was decreased by 6.5mmHg and diastolic blood pressure (DBP) was decreased by 4.6mmHg.

Traditional physician-led services are usually focused on the medical management of hypertension. However, as part of a holistic approach, counselling and education interventions are considered an essential supplement to medical management, and nurses play a key role in patient education, medication management, and chronic disease monitoring. Nurses can provide timely follow-up, track patient progress, and offer guidance on medication adherence and lifestyle changes, which are crucial for hypertension control.

Rationale/Justification:

According to STEPS survey 2019 in Nepal, 24.5% of adults were hypertensive, with 47.3% unaware of their condition, 29.6% of those with hypertension were receiving treatment and among those receiving treatment, only 14.8% had their blood pressure under control. Hypertension control in Nepal faces significant challenges due to limited access to health facilities, particularly in rural areas which are due to geographical constraints and shortage of healthcare personnel which are compounded by low public awareness and inadequate follow up. Hypertension, sometimes called the ''disease of habit,'' can be prevented and managed through adequate lifestyle adjustments. Nurse-led telehealth interventions are helpful in overcoming the geographical barriers and increasing expert care without the need for extensive travel and also benefit patients from improved communication and care coordination. Studies have suggested that nurse-led telehealth decreases the SBP and DBP.

However, evidence regarding telehealth for hypertension control and nurse-led telehealth in low-middle income countries, particularly Nepal is limited. As the burden of uncontrolled hypertension is high, this study aims to evaluate the effectiveness of a nurse-led telehealth intervention compared to standard care in improving hypertension control among individuals with hypertension in Nepal.

General Objectives:

To evaluate the effectiveness of nurse-led telehealth in primary care for hypertension control in Nepal.

Specific Objective:

Evaluate the effectiveness of nurse-led telehealth compared to standard care in reducing systolic blood pressure among individuals with hypertension over six months.

Research Hypothesis There is no significant difference in the systolic BP between individuals with hypertension who received nurse-led telehealth compared to those who received standard of care.

Study Variables

Dependent variables:

Primary: Systolic blood pressure; Secondary: Diastolic blood pressure, blood pressure control, Medication adherence, Hypertension selfcare, acceptability, appropriateness and feasibility of nurse-led telehealth Independent variables: Nurse-led telehealth Socio-demographic and clinical variables: Age, gender, education level, ethnicity, marital status, religion, occupation, BMI, socioeconomic status, family type, salt intake, smoking, alcohol intake, physical activity, Family history of Hypertension, duration of Hypertension, number of anti-hypertensive drugs, distance to nearby health service, frequency of follow-up visits, medical insurance, comorbidity Research Design: Randomized controlled trial

Number of participants and Justification:

A sample size of 294 patients per group is required in order to have 80% power to detect a difference in SBP of 5 mm Hg between intervention and control groups, with an assumption of SD 21.63 mm Hg, based on the findings from the study19 Allowing for a 20% participant drop out, we will seek to recruit 353 participants in each group resulting in a total sample size of 706 participants.

Study Population:

Individuals with hypertension aged 30 years and above residing at Panchkhal and Panauti Municipality meeting the inclusion criteria.

Sampling Unit:

Adults aged 18 years and above who meet the specified inclusion criteria and who provide consent for the study participation.

Data Collection technique:

In this study, The Investigators will recruit patients directly from the community in selected wards of Panchkhal and Panauti Municipalities. I along with 1 Medical Officer and few research nurses will conduct a series of hypertension screening camp in collaboration with local health Offices and Female Health Volunteers to identify individuals with elevated blood pressure or diagnosed hypertension. On the first day, The Investigators measure at least two blood pressure measurement of individual participants will be taken in the left arm in the sitting position after 5 min rest with a validated electronic automated sphygmomanometer, 3 reading spaced 1-2 min apart and the average value of second and third reading will be used for diagnosis. If the patients have elevated readings (>140/90 mmHg), we will ask them to return the next day for a repeat measurement (For newly Diagnosed). If a participant's BP remains high on both days, we will confirm them as hypertensive and consider for recruitment. We will also recruit the patients who have high BP and are already diagnosed with hypertension or those who are normotensive but currently on antihypertensive medication for the study. We will prepare a list of eligible individuals and contact for informed consent and study enrollment.

Randomization Sequence generation: Participants who meet the eligibility criteria after screening will be randomly assigned to either the intervention group or the control group on the basis of computer-generated random sequence using Stata 14. Someone independent of the research team will generate the sequence Allocation concealment: The randomization sequence will be placed in sealed envelopes and are opened sequentially only after the participants are recruited.

Implementation: An independent statistician will generate the random allocation sequence using computer-based randomization software with a 1:1 allocation ratio. Research nurses will be responsible for screening participants, obtaining informed consent, and enrolling eligible participants into the study.

Blinding: None of the study participants will be blinded to group allocation because both the participants and nurses will know who is receiving the telehealth intervention as it involves direct interaction.

Data collection tools:

For baseline assessment, the Investigators will use structured interview questionnaires for sociodemographic and clinical variables like Age, gender, education level, ethnicity, marital status, religion, occupation, BMI, socioeconomic status, family type, smoking, alcohol intake, physical activity, Family history of Hypertension, duration of Hypertension, Number of anti-hypertensive drugs, frequency of follow-up visits, medical insurance, distance to nearby health service, comorbidity; Hypertension Self Care will be measured by using Hypertension Selfcare profile developed by Han et.al. translated in Nepali language by the author for use in this study, Medication adherence using Hill-Bone Compliance to High Blood Pressure Therapy Scale (HBCTS) developed by Kim et al21 and translated and validated into Nepalese version by Shakya et al.22 Physical Activity will be measured using the Global Physical Activity Questionnaire by World Health Organization23 and translated and validated into Nepali version by Algallai et.al.24 Blood pressure will be measured using a validated automated digital BP monitor (Omron HEM-7121). Participants' height will be measured using a portable stadiometer to the nearest 0.1 cm, and weight will be recorded using a calibrated digital scale to the nearest Plan for data analysis

Descriptive data analysis:

The Investigators will present the descriptive analysis for baseline characteristics comparing the intervention and usual care group as frequency (percentage) for categorical variables whereas the mean (SD) for normally distributed continuous variables and median (IQR) for skewed variables.

Primary analysis: The Investigators will conduct the primary analysis according to the intent-to-treat principle comparing differences in mean SBP (net change in mean SBP from baseline to 6 months follow-up) between the intervention and control group. The Investigators will utilize univariate linear regression models with intervention status (yes/no) as independent variables and systolic blood pressure as outcome.

Secondary analysis: If participants do not receive the intervention after randomization, the investigator will conduct a per-protocol analysis excluding these individuals. In this analysis, the investigators will adjust for potential confounding variables such as baseline systolic and diastolic blood pressure, blood pressure control status, medication adherence, hypertension self-care, as well as relevant socio-demographic and clinical characteristics.

Expected outcome of the research results:

The expected clinical outcomes of this study include a significant reduction in systolic and diastolic blood pressure, and an increased proportion of participants achieving controlled blood pressure. The intervention is accepted to be perceived as acceptable, appropriate and feasible by both patients and nurses. The expected behavioral outcomes are improved medication adherence and enhanced hypertension self-care practices. If nurse-led intervention proves effective, it could serve as a scalable and sustainable model for hypertension management in low-resource settings where access to specialists is limited.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30 years and above
* Blood pressure at baseline of more than 140 or 90 mm Hg on at least two separate visits or under antihypertensive medications
* Willing to monitor their blood pressure and self-titrate medication
* Possess a smartphone with internet access and WhatsApp/Viber at least biweekly
* No cognitive deficit and able to communicate effectively to carry out study tasks
* Not planning to change residence during the 6-month follow-up

Exclusion Criteria:

* Pregnant women
* Patients in hypertensive crisis (BP ≥180/120 mm Hg)
* Had a stroke in the past 30 days or are on dialysis
* Individuals with self-reported serious advanced illness such as terminal cancer
* Patients enrolled in other BP research during the same period

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure | 6 months
  It is the difference in Systolic Blood Pressure from the endline to baseline measured in mmHg.

SECONDARY OUTCOMES:
Change in Diastolic Blood pressure | 6 months
  It is the difference in Systolic Blood Pressure from the endline to baseline measured in mmHg.
Blood pressure control | 6 months
  It is the difference in blood pressure control from the endline to baseline measured in percentage.
Medication Adherence | 6 months
  it is the difference in Medication Adherence measured using Hill-Bone Compliance to High Blood Pressure Therapy Scale (HBCTS) from endline to baseline.
Hypertension selfcare | 6 months
  It is the difference in the Hypertension selfcare measured by using Hypertension Selfcare profile from endline to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Archana Shrestha, PhD, Principal Investigator — Kathmandu University School of Medical Sciences
Locations (1):
- Kathmandu University School of Medical Sciences, Dhulikhel, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bulto LN, Roseleur J, Noonan S, Pinero de Plaza MA, Champion S, Dafny HA, Pearson V, Nesbitt K, Gebremichael LG, Beleigoli A, Gulyani A, Schultz T, Hines S, Clark RA, Hendriks JM. Effectiveness of nurse-led interventions versus usual care to manage hypertension and lifestyle behaviour: a systematic review and meta-analysis. Eur J Cardiovasc Nurs. 2024 Jan 12;23(1):21-32. doi: 10.1093/eurjcn/zvad040. PMID 37130339
- [Background] Omboni S, McManus RJ, Bosworth HB, Chappell LC, Green BB, Kario K, Logan AG, Magid DJ, Mckinstry B, Margolis KL, Parati G, Wakefield BJ. Evidence and Recommendations on the Use of Telemedicine for the Management of Arterial Hypertension: An International Expert Position Paper. Hypertension. 2020 Nov;76(5):1368-1383. doi: 10.1161/HYPERTENSIONAHA.120.15873. Epub 2020 Sep 14. PMID 32921195
- [Background] McManus RJ, Little P, Stuart B, Morton K, Raftery J, Kelly J, Bradbury K, Zhang J, Zhu S, Murray E, May CR, Mair FS, Michie S, Smith P, Band R, Ogburn E, Allen J, Rice C, Nuttall J, Williams B, Yardley L; HOME BP investigators. Home and Online Management and Evaluation of Blood Pressure (HOME BP) using a digital intervention in poorly controlled hypertension: randomised controlled trial. BMJ. 2021 Jan 19;372:m4858. doi: 10.1136/bmj.m4858. PMID 33468518
- See also: Home and Online Management and Evaluation of Blood Pressure (HOME BP) using a digital intervention in poorly controlled hypertension: randomised controlled trial. — https://www.bmj.com/content/372/bmj.m4858
- See also: Effectiveness and acceptability of a mobile phone text messaging intervention to improve blood pressure control (TEXT4BP) among patients with hypertension in Nepal: A feasibility randomised controlled trial. — https://pubmed.ncbi.nlm.nih.gov/35342691/
- See also: Effectiveness of nurse-led interventions versus usual care to manage hypertension and lifestyle behaviour: a systematic review and meta-analysis. — https://pubmed.ncbi.nlm.nih.gov/37130339/